CLINICAL TRIAL: NCT04339790
Title: Mental Health Impact of COVID-19 Pandemic on NIMH Research Participants and Volunteers
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999920085; 20-M-N085
Record Dates: First submitted 2020-04-08; First posted 2020-04-09 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-04-12

CONDITIONS: Healthy Volunteer; Mood Disorder; Anxiety Disorder; Preexisting Medical Condition
Keywords: Coronavirus; COVID-19; Mental Health; Environmental Stressor; Distress; Natural History
MeSH Terms: conditions — Mood Disorders; Anxiety Disorders; Coronavirus Infections; COVID-19; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- New study participant: Individuals who respond to study website or advertisements for the study who have not previously been a NIMH study participant
- NIMH Study Participant: Individuals who have previously consented for a NIMH study

SUMMARY:
Background:

The COVID-19 outbreak has caused many changes to people s normal social patterns. The respiratory illness has been the major focus of public health efforts. But most experts also agree that government and public health mandates to slow the spread of the illness, such as social distancing, have a significant effect on people s mental health. Environmental stressors, such as constraints on activities, social contact, and access to resources, take a toll. Researchers want to learn how stressors related to COVID-19 affect mental health over time.

Objective: To learn the relationship between stressors related to COVID-19 and self-rated measures of mental health symptoms and distress among a range of people.

Eligibility:

English-speaking adults ages 18 and older

Design:

This study will be conducted online.

Participants will give their first and last name and email address. They will indicate if they have ever been in an NIH research study. They will get a username and password.

Every 2 weeks for up to 6 months, participants will complete online study surveys. They will get email reminders. Some surveys will be repeated. At the end of the study, they will complete a set of end-of-study surveys.

The surveys will ask about the following:

Age, sex, race, and other sociodemographic data

Mental and medical illness history and treatment

Family medical history

Mobility, self-care, and life activities

Behaviors related to alcohol and substance use disorder

Mental illness symptoms

Psychological distress

Stressors caused by the COVID-19 pandemic.

Participants will get links to mental health resources, such as hotlines. They will also get guidance on steps to take to seek care or support.

Study website: nimhcovidstudy.ctss.nih.gov

DETAILED DESCRIPTION:
Study Description: This protocol leverages existing NIMH studies and participants to accomplish time-sensitive research on the mental health impact of environmental stressors imposed by the COVID-19 pandemic. The study will describe the relationship between stressors related to COVID-19 and self-rated measures of mental health symptoms and distress among a range of participants including various patient populations and healthy volunteers. The utilization of a study website to consent and survey participants online is an efficient and timely way to collect research data during this unique public health crisis.

Objectives: The primary objective is to describe the relationship between stressors related to COVID-19 and self-rated measures of mental health symptoms and distress among a range of participants including various patient populations and healthy volunteers. The secondary objectives are to determine whether existing mental health concerns moderates this relationship and to identify risk and resilience factors among study participants regarding the mental health impact of the COVID-19 pandemic.

Endpoints: The primary endpoints are descriptive data on stressors experienced as a result of the COVID-19 pandemic, and emotional, behavioral, and clinical symptoms. These endpoints will be measured repeatedly using an online platform for up to 6 months. These repeated measures will be combined with previously collected phenotype data on NIMH participants as allowed.

Study Population: The sample size will be up to 10,000 and will include participants 18 years and older of both sexes, any gender, and health status. They must be English-speaking. The study population will include patient and volunteer participants who have consented for a NIMH study in the past as well as new participants from the general population who respond to advertisements for the NIMH COVID study but who have not previously been a NIMH study participant. The NIMH COVID study participants may or may not be local to the Metropolitan Washington DC area but since the study will be conducted entirely online, this is not relevant.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* 18 years of age and older.
* Able to read and write English.
* Able to provide informed consent online using study website.

EXCLUSION CRITERIA:

There are no exclusion criteria for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population for the NIMH COVID study will include patient and volunteer participants who have consented for a NIMH study in the past as well as new participants from the general population whorespond to advertisements for the NIMH COVID study but who have not previously been a NIMH studyparticipant. The NIMH COVID study participants may or may not be local to the Metropolitan WashingtonDC area but since the study will be conducted entirely online, this is not relevant.
Sampling Method: Non-Probability Sample
Enrollment: 3655 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-06-02 (Actual)

PRIMARY OUTCOMES:
NIMH COVID Study survey - adult responses | Biweekly online responses
  Thoughts and feelings about mental health impact of COVID-19

SECONDARY OUTCOMES:
DSM XC and KS survey | Biweekly online self report
  Ratings on measures of mental health symptoms and distress

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Y Chung, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Cohen S, Gianaros PJ, Manuck SB. A Stage Model of Stress and Disease. Perspect Psychol Sci. 2016 Jul;11(4):456-63. doi: 10.1177/1745691616646305. PMID 27474134
- [Background] Kendler KS, Hettema JM, Butera F, Gardner CO, Prescott CA. Life event dimensions of loss, humiliation, entrapment, and danger in the prediction of onsets of major depression and generalized anxiety. Arch Gen Psychiatry. 2003 Aug;60(8):789-96. doi: 10.1001/archpsyc.60.8.789. PMID 12912762
- [Derived] Gibbons AB, Farmer C, Shaw JS, Chung JY. Examining the factor structure of the DSM-5 Level 1 cross-cutting symptom measure. Int J Methods Psychiatr Res. 2023 Jun;32(2):e1953. doi: 10.1002/mpr.1953. Epub 2022 Nov 1. PMID 36318494